CLINICAL TRIAL: NCT02390401
Title: Incisional VAC at Cesarean Section for Prevention of Post Operative Wound Complications in the Obese
Brief Title: Vacuum Assisted Closure for Cesarean Section
Acronym: VACCS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Continuation was futile per calculation recommend by data & safety monitoring committee
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Southern New Hampshire Medical Center (Other)
Responsible Party: Principal Investigator, Zachary Spalding, Physician-Resident, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D15054
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vacuum-assisted closure (VAC) (Experimental): Prevena (VAC) device
  Interventions: Device: Vacuum-assisted closure
- Standard sterile dressing (Active Comparator): Standard sterile dressing
  Interventions: Device: Standard sterile dressing

INTERVENTIONS:
Device: Vacuum-assisted closure — Prevena (VAC) device at the time of primary closure for a cesarean section, left in place for 5-7 days postoperatively.
  Other Names: Prevena; Incisional VAC
  Arms: Vacuum-assisted closure (VAC)
Device: Standard sterile dressing — Standard sterile dressing at the time of primary closure for a cesarean section, left in place for 1-2 days postoperatively.
  Arms: Standard sterile dressing

SUMMARY:
To study if incisional vacuum-assisted closure can decrease the risk of infection in cesarean section incisions in the obese compared with standard sterile dressing.

DETAILED DESCRIPTION:
The prevalence of obesity (defined as body mass index (BMI, kg/m2) ≥ 30) has significantly increased, affecting approximately 35% of adult females in the United States, according to CDC 2009-2010 statistics. Obesity has a significant impact on pregnancy, including increased need for cesarean section and post-operative wound complications. Infection rates have been reported to be between 10 and 30%. The advent in 1997 of negative pressure therapy (NPT), also known as vacuum assisted closure (VAC), has vastly changed wound care management. Briefly, VAC has been traditionally applied to a chronic wound to create negative or sub-atmospheric pressure, thus promoting wound healing by decreasing edema and increasing blood flow and formation of granulation tissue. Use of this therapy at the time of primary closure of a surgical incision (first trialed in 2006 and termed "Incisional VAC") has provided a promising approach to reducing post-operative wound infection. Incisional VAC has been explored primarily in the orthopedic and cardiothoracic fields, but very few studies have examined the use on abdominal incisions, and only one to date on cesarean section incisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone cesarean section for delivery; have a BMI greater or equal to 35. All cases of cesarean section including primary and repeat, scheduled and urgent.

Exclusion Criteria:

* Patients who deliver vaginally; age less than 18 years old; silver allergy; non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Post-operative wound infection | 6 weeks post-operative
  Determine number of post-operative wound infections

SECONDARY OUTCOMES:
Rate of seroma | 6 weeks post-operative
  Calculate incidence of seroma
Rate of hematoma | 6 weeks post-operative
  Calculate incidence of hematoma
Deep and superficial infection | 6 weeks post-operative
  Calculate incidence of deep and superficial infection
Readmission for infection | 6 weeks post-operative
  Calculate incidence of readmission to hospital for infection due to cesarean incision
Re-operation | 6 weeks post-operative
  Calculate incidence of re-operation to patients enrolled in study
Antibiotic treatment | 6 weeks post-operative
  Calculate incidence of need for antibiotic treatment for enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Spalding, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Kristina Wihbey, MD, Study Chair — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Women's Care of Nashua, Nashua, New Hampshire
  - Dartmouth-Hitchcock Nashua, Nashua, New Hampshire
  - Southern New Hampshire Medical Center, Nashua, New Hampshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wihbey KA, Joyce EM, Spalding ZT, Jones HJ, MacKenzie TA, Evans RH, Fung JL, Goldman MB, Erekson E. Prophylactic Negative Pressure Wound Therapy and Wound Complication After Cesarean Delivery in Women With Class II or III Obesity: A Randomized Controlled Trial. Obstet Gynecol. 2018 Aug;132(2):377-384. doi: 10.1097/AOG.0000000000002744. PMID 29995726